CLINICAL TRIAL: NCT05726552
Title: Effect of Laughter Therapy on Hemodialysis Patients: A Randomized Controlled Study
Brief Title: The Effect of Laughter Therapy on Hemodialysis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zonguldak Bulent Ecevit University (Other)
Collaborators: Marmara University (Other)
Responsible Party: Principal Investigator, Canan Eraydın, Lecturer, Zonguldak Bulent Ecevit University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: ZNGLDKBEUSBF
Record Dates: First submitted 2023-01-24; First posted 2023-02-14 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Laughter Therapy; Depression, Anxiety; Hemodialysis; Life Quality
MeSH Terms: conditions — Depression; Anxiety Disorders | interventions — Laughter Therapy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Only the statistical analyst (outcome assessor) was blinded to group allocation. Participants and investigators were aware of the intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laughter Therapy group (Experimental): Hemodialysis patients(40) enrolled in the laughter therapy group will receive a total of 12 sessions of laughter therapy, 50 minutes, 3 days a week.
  Interventions: Other: Laughter therapy
- Control (No Intervention): No attempt will be made to hemodialysis patients in this group.

INTERVENTIONS:
Other: Laughter therapy — Laughter therapy will be applied for 50 minutes, 12 sessions, 3 days a week. The therapy, which starts with the stimulation of the acupuncture points in the palm and acquaintance with hand clapping for an average of 10 minutes, continues with deep breathing and breathing exercises that include diaphragmatic breathing. The childish games section, which is played to reveal and trigger simulated laughter, is the section where laughter starts as "if" and turns into reality.
  The last part is the part where the group makes eye contact for no reason and for no reason, and laughs for at least 3 minutes unconditionally. In the last part, wish meditation and relaxation sessions are performed.
  Arms: Laughter Therapy group

SUMMARY:
Internet-based behavioral therapy applications made during the quarantine and isolation period during the pandemic process, and the application of laughter therapy, which is a group-oriented technique that increases the feeling of togetherness and happiness, can be used as an online method to reach large masses. However, since there are a limited number of studies in the literature on online laughter therapy in patients and not all sessions are online in the study, it was thought that more and methodological studies are needed to confirm the effectiveness of the therapy on the applicability of the online platform. Therefore, this study was conducted to evaluate the blood cortisol levels, depression, anxiety, stress levels and quality of life of laughter therapy in hemodialysis patients.

DETAILED DESCRIPTION:
In this research, laughter therapy applied to hemodialysis patients; This is an experimental design with pretest and posttest control groups in order to examine the effects on serum cortisol levels, depression, anxiety, stress levels and quality of life. The study will be conducted between April 2021 and September 2022 on 80 patients who are receiving hemodialysis treatment in two Dialysis Centers in Zonguldak city center and meet the inclusion criteria. Introductory information form, Depression Anxiety and Stress Scale, Kidney Disease Quality of Life Form will be used in the study and blood samples will be taken from the patients for cortisol. Laughter therapy will be applied three days a week, for a total of 12 sessions for 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Do not prevent you from doing laughter yoga (having undergone abdominal surgery in the last three months, uncontrollable hypertension, chronic cough, incontinence, acute low back pain, acute mental disorders, consumption of antipsychotic drugs, glaucoma, hernia, epilepsy)
* History of psychiatric illness (major depression, alcohol abuse, substance abuse, schizophrenia or paranoid disorders, personality disorder, somatoform disorder)
* Standardized Mini Mental Test (SMMT) score 24>
* Not doing laughter yoga before
* Being able to use smart phone/computer/tablet and using internet applications actively

Exclusion Criteria:

* Initiation of medication that may affect serum cortisol levels
* Diagnosis of psychiatric illness during sessions
* Surgery on the abdominal region during laughter sessions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2022-09-25 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
Kidney Disease Quality of Life Scoring | 4 months
  The Kidney Disease Quality of Life Scale (KDQOL-SF) is a scale used to evaluate the well-being and function of individuals with kidney disease and undergoing dialysis treatment. The scale was developed by Hays et al. in the USA in 1994 (Hays et al., 1994). The validity and reliability study in our country was carried out by Yıldırım et al. in 2007.

SECONDARY OUTCOMES:
Cortisol level | 4 months
  All cortisol levels before and after laughter were measured in a fully automatic Roche Cobas 8000 device using the elecsys cortisol II kit, according to the electrochemiluminescence immunoassay method in the central laboratory of a State Hospital.
Depression, Anxiety, Stress scale | 4 months
  Description: Depression Anxiety Stress Scale (DASS-21) was first developed by Lovibond (1995) as 42 items. The adaptation of the 21-question DASS scale used in the study was made by Henry and Crawford (2005), and it was revealed that the short form could be used. The scale, which was revised by Henry and Crawford, was adapted into Turkish by Yılmaz et al. (2017). In this scale, there are 7 questions each to measure the dimensions of depression, anxiety and stress. The first 7 questions on the scale are about anxiety, 7 questions between 8-14 are about depression and 7 questions between 15-21 are about stress. The scale has a 4-point Likert-type rating of 0 "not at all suitable for me", 1 "somewhat appropriate for me", 2 "usually suitable for me", and 3 "completely suitable for me". Cronbach Alpha value for each sub-dimension of the adapted scale; Anxiety (7 items) 0.80; It was found to be 0.81 for Depression (7 items) and 0.75 for Stress (7 items).

CONTACTS AND LOCATIONS:
Overall Officials: Şule ECEVİT ALPAR, Doctorate, Study Director — Marmara University
Locations (1):
- Zonguldak Bülent Ecevit University, Zonguldak, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kim J, Yun KS, Cho A, Kim DH, Lee YK, Choi MJ, & Park HC. High cortisol levels are associated with oxidative stress and mortality in maintenance hemodialysis patients. BMC nephrology, 2022; 23(1), 1-9. Ko Y, Lee ES, & Park S. Effects of laughter therapy on the stress response of married immigrant women in South Korea: A randomized controlled trial. Health Care Women Int. 2022;43(5): 518-531. 112. Ko YJ, Hyun MY. Effects of laughter therapy on pain, depression, and quality of life of elderly people with osteoarthritis. J Korean Acad Psychiatr Ment Health Nurs. 2013; 22(4): 359-67.
- [Result] Aminoff V, Sellen M, Sorliden E, Ludvigsson M, Berg M, Andersson G. Internet-Based Cognitive Behavioral Therapy for Psychological Distress Associated With the COVID-19 Pandemic: A Pilot Randomized Controlled Trial. Front Psychol. 2021 Jun 14;12:684540. doi: 10.3389/fpsyg.2021.684540. eCollection 2021. PMID 34194374
- [Result] Eraydin C, Alpar SE. The effect of laughter therapy on nursing students' anxiety, satisfaction with life, and psychological well-being during the COVID-19 pandemic: Randomized controlled study. Adv Integr Med. 2022 Sep;9(3):173-179. doi: 10.1016/j.aimed.2022.06.006. Epub 2022 Jun 24. PMID 35782290